CLINICAL TRIAL: NCT06753032
Title: Impact of Positive & Negative Lens-Induced Defocus on Contrast-Sensitivity in Myopic & Non-Myopic Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MSRSW/Batch-Fall22/750
Record Dates: First submitted 2024-12-13; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- interventional group (Experimental)
  Interventions: Diagnostic Test: Positive Lens-Induced Defocus Using Spectacle Lenses (+2.00 D) for Myopic Participants
- Interventional group II (Experimental)
  Interventions: Diagnostic Test: Negative Lens-Induced Defocus Using Spectacle Lenses (-2.00 D) for Myopic Participants
- Interventional group III (Active Comparator)
  Interventions: Combination Product: Positive Lens-Induced Defocus Using Spectacle Lenses (+2.00 D) for Non-Myopic Participants
- Interventional group IV (Active Comparator)
  Interventions: Combination Product: Negative Lens-Induced Defocus Using Spectacle Lenses (-2.00 D) for Non-Myopic Participants

INTERVENTIONS:
Diagnostic Test: Positive Lens-Induced Defocus Using Spectacle Lenses (+2.00 D) for Myopic Participants — Intervention Description: This group will be exposed to positive defocus induced by +2.00 D spectacle lenses. The lenses are designed to create optical blur to evaluate the effects on contrast sensitivity and visual fatigue. Measurements will be conducted at baseline, 2 weeks, and 4 weeks after exposure to assess changes in visual function."
  Arms: interventional group
Diagnostic Test: Negative Lens-Induced Defocus Using Spectacle Lenses (-2.00 D) for Myopic Participants — Intervention Description: This group will be exposed to negative defocus induced by -2.00 D spectacle lenses. The induced defocus will allow for the evaluation of its impact on contrast sensitivity and visual fatigue. Assessments will be carried out at baseline, 2 weeks, and 4 weeks."
  Arms: Interventional group II
Combination Product: Positive Lens-Induced Defocus Using Spectacle Lenses (+2.00 D) for Non-Myopic Participants — ntervention Description: This group will undergo positive defocus using +2.00 D spectacle lenses. The intervention aims to examine the effect of induced defocus on contrast sensitivity and visual fatigue in non-myopic participants. Data will be collected at baseline, 2 weeks, and 4 weeks."
  Arms: Interventional group III
Combination Product: Negative Lens-Induced Defocus Using Spectacle Lenses (-2.00 D) for Non-Myopic Participants — Intervention Description: This group will experience negative defocus induced by -2.00 D spectacle lenses. The purpose is to evaluate how negative lens-induced defocus affects contrast sensitivity and visual fatigue in non-myopic participants. Measurements will be taken at baseline, 2 weeks, and 4 weeks.
  Arms: Interventional group IV

SUMMARY:
examines the influence of lens-induced defocus on contrast sensitivity-a crucial aspect of visual performance.Each participant experiences both positive and negative defocus through different lenses, with measurements taken for contrast sensitivity using the Pelli-Robson chart. Outcomes are evaluated at baseline, 2 weeks, and 4 weeks to understand the effect of defocus over time.

DETAILED DESCRIPTION:
Additional data on symptoms like visual fatigue and computer vision syndrome are gathered using the Visual Fatigue Questionnaire (VFQ) and the Computer Vision Syndrome Questionnaire (CVS-Q), respectively. This study's findings could be instrumental in refining optical treatments, offering insights into how defocus impacts visual function across refractive conditions. Results may ultimately benefit optometric practices by guiding lens prescriptions for improved contrast sensitivity and quality of life for myopic and non-myopic individuals alike.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 50 years.
* Participants with a confirmed diagnosis of myopia or non-myopia.
* Best corrected visual acuity of 20/30 or better.
* No history of ocular surgery or significant ocular disease.
* Informed consent was obtained.

Exclusion Criteria:

* Individuals with a history of systemic diseases affecting vision (e.g., diabetes, hypertension).
* Presence of binocular vision anomalies or strabismus.
* Pregnant or nursing women.
* Any current use of medications affecting visual function (e.g., medications causing visual side effects).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-02-28 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Contrast Sensitivity | 12 Months
  Measured with the Pelli-Robson Contrast Sensitivity Chart, capturing changes in participants' ability to detect low-contrast visual stimuli under defocus conditions.
Visual Fatigue | 12 months
  Evaluated with the Visual Fatigue Questionnaire (VFQ) and Computer Vision Syndrome assessing symptoms like eye strain, discomfort, and fatigue following lens-induced defocus.

CONTACTS AND LOCATIONS:
Locations (1):
- Tehsil Headquarters (THQ), Taunsa, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No